CLINICAL TRIAL: NCT01582607
Title: Intrathecal Plain Bupivacaine, Ropivacaine and Levo-bupivacaine With or Without Fentanyl for Elective c Section.
Brief Title: Subarachnoid Administration of Levobupivacaine for Cesarean Section
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Nikolaos G. Flaris, Anesthesiologist,MD, University of Patras
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 3089
Record Dates: First submitted 2012-04-14; First posted 2012-04-20 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Stillborn Caesarean Section
MeSH Terms: interventions — Bupivacaine; Ropivacaine; Levobupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Group B (Active Comparator): subarachnoid administration of 2.0 mL (10mg) plain bupivacaine hydrochloride 0.5%
  Interventions: Drug: Bupivacaine plain
- Group R (Active Comparator): subarachnoid administration of 2.0 ml (15mg) plain ropivacaine 0.75%
  Interventions: Drug: Ropivacaine plain
- Group LB (Active Comparator): subarachnoid administration of 2.0 ml (10mg) plain levo-bupivacaine hydrochloride 0.5%
  Interventions: Drug: Levobupivacaine plain
- Group RF (Active Comparator): subarachnoid administration of 2.0 ml (15mg) plain ropivacaine 0.75% with 0.2 ml (10 μg) fentanyl
  Interventions: Drug: ropivacaine plain +. fentanyl
- Group BF (Active Comparator): subarachnoid administration of 2.0 ml (10mg) plain bupivacaine 0.5% with 0.2 ml (10 μg) fentanyl
  Interventions: Drug: bupivacaine plain +fentanyl
- Group LBF (Active Comparator): subarachnoid administration of 2.0 ml (10mg) plain levo-bupivacaine 0.5% with 0.2 ml (10 μg) fentanyl
  Interventions: Drug: Levobupivacaine plain +fentanyl

INTERVENTIONS:
Drug: Bupivacaine plain — 2.0 mL (10mg) plain bupivacaine hydrochloride 0.5% intrathecally
  Other Names: Marcaine Spinal 5 mg/ml, AstraZeneca
  Arms: Group B
Drug: Ropivacaine plain — 2.0 ml (15mg) plain ropivacaine 0.75% intrathecally
  Other Names: Naropeine 7.5mg/ml, AstraZeneca
  Arms: Group R
Drug: Levobupivacaine plain — 2.0 ml (10mg) plain levo-bupivacaine hydrochloride 0.5% intrathecally
  Other Names: Chirocaine 5mg/ml, Abbott Laboratories
  Arms: Group LB
Drug: bupivacaine plain +fentanyl — 2.0 ml (10mg) plain bupivacaine 0.5% with 0.2 ml (10 μg) fentanyl intrathecally
  Other Names: Marcaine Spinal 5 mg/ml; Fentanyl, 50μg/ml, Janssen-Cilag, Belgium
  Arms: Group BF
Drug: ropivacaine plain +. fentanyl — 2.0 ml (15mg) plain ropivacaine 0.75% with 0.2 ml (10 μg) fentanyl intrathecally
  Other Names: Naropeine 7.5mg/ml, AstraZeneca; Fentanyl, 50μg/ml, Janssen-Cilag, Belgium
  Arms: Group RF
Drug: Levobupivacaine plain +fentanyl — 2.0 ml (10mg) plain levo-bupivacaine 0.5% with 0.2 ml (10 μg) fentanyl intrathecally
  Other Names: Chirocaine 5mg/ml, Abbott laboratories; Fentanyl, 50μg/ml, Janssen-Cilag, Belgium
  Arms: Group LBF

SUMMARY:
The purpose of the investigators study is to compare the clinical effects and side-effects of these three local anaesthetics as sole agents or with the supplementation with fentanyl for c-section, especially when administered in doses achieving approximately an ED 50.

DETAILED DESCRIPTION:
Intrathecal (i.t.) administration of isobaric bupivacaine, ropivacaine and levobupivacaine with or without addition of fentanyl for c-section do not exist to date .

Parturients scheduled for elective caesarean section will be allocated to receive double-blindly i.t. isobaric bupivacaine 10 mg, ropivacaine 15mg , levobupivacaine 10mg or the same local anaesthetics with 10 μg fentanyl respectively. Sensory block (pin prick test) and motor block (Bromage scale) profile, intraoperative and postoperative analgesia, haemodynamics and side effects will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Parturients scheduled for elective c section
* Stillborn
* Normal cardiotocogram

Exclusion Criteria:

* BMI>35kg/m2
* Height <150cm or >185cm
* Age (<18, >40)
* ASA > II
* Multiple gestation
* Pregnancy complications (eclampsia, GDP, placenta previa, >2 previous c section)
* Contraindication to spinal anaesthesia
* Failure to educate the patient, language barrier
* Patient preferred GA

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-04 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Sensory block | up to 150 minutes average
  sensory block (pin prick test): every 1 min until 30min, every 5 min until 60min. every 10 min until regression to O1 (average 150 minutes)
Motor block | up to 150 minutes
  Motor block (Bromage scale): every 1 min until 30min, every 5 min until 60min. every 10 min until complete recovery of motor function (average 150 minutes)

SECONDARY OUTCOMES:
Hemodynamics profile (arterial pressure. heart rate) | up to 150 minutes average
  Measurement of arterial pressure and heart rate every 1 min for the first 30 min, every 5 min until 60 min, every 10 min until regression of sensory or motor block(average 150 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos G Flaris, MD, Principal Investigator — University Hospital of Patras; Kriton S Filos, Professor, Study Director — University Hospital of Patras
Locations (1):
- University Hospital of Patras, Department of Anesthesiology, Pátrai, Achaia, Greece